CLINICAL TRIAL: NCT05463809
Title: A Randomized Controlled Trial of Continuous Gastrocnemius Plane Block and Intravenous Analgesia After Foot and Ankle Surgery
Brief Title: Compare Continuous Gastrocnemius Plane Block With Intravenous Analgesia After Foot and Ankle Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Han Liu
Record Dates: First submitted 2022-07-04; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Foot Ankle Injuries
Keywords: nerve block; Continuous Gastrocnemius plane block
MeSH Terms: interventions — Ropivacaine; Oxycodone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Ropivacaine-controlled analgesia pump (Experimental): A single injection of 0.375% Ropivacaine 15 milliliters was given into the common peroneal nerve, medial sural cutaneous nerve, and lateral sural cutaneous nerve. Than，a catheter was placed in the gastrocnemius plane, and a 0.125% ropivacaine-controlled analgesic pump was applied.(The formulation was 0.125% ropivacaine at 300 milliliters, with a background dose of 3 milliliters/hours, a patient-controlled analgesia(PCA) dose of 8 milliliters, and a locking time of 25 minutes.）
  Interventions: Drug: Continuous Gastrocnemius plane block with ropivacaine
- Control group: oxycodone-controlled analgesia pump (Experimental): No treatment was given preoperatively, and postoperative oxycodone patient-controlled intravenous analgesia(PCIA). After awakening, intravenous oxycodone was titrated according to numerical rating scale(NRS) score, providing analgesia without background dose of oxycodone patient-controlled intravenous analgesia(PCIA) pump (single dose 1 milligram, locking time 5 minutes, 14 hours limit 12 milligrams)
  Interventions: Drug: oxycodone

INTERVENTIONS:
Drug: Continuous Gastrocnemius plane block with ropivacaine — After extubation, the patient was routinely monitored for his vital signs.The nerve block operation was performed by the same doctor: let the patient take the lateral decubitus position, use the ultrasonic high-frequency array probe under the popliteal socket to scan the sciatic nerve, move the probe down to find the tibial nerve and the common peroneal nerve, and then a single injection of 0.375% Ropivacaine 15milliliters was given into the common peroneal nerve, medial sural cutaneous nerve, and lateral sural cutaneous nerve. Then avoid common peroneal nerve, use the indwelling needle (16GA 3.25 IN), and put the catheter after saline expansion.
  Other Names: Automatic analgesic pump
  Arms: Experimental group: Ropivacaine-controlled analgesia pump
Drug: oxycodone — The patient was revived and received intravenous oxycodone titration according to the numerical rating scale (NRS) score, and was treated with no background dose of oxycodone patient-controlled intravenous analgesia (PCIA) pump for analgesia.
  Other Names: Automatic analgesic pump
  Arms: Control group: oxycodone-controlled analgesia pump

SUMMARY:
This study aims to evaluate the efficacy and safety of a continuous gastrocnemius plane block for perioperative analgesia in patients undergoing foot and ankle surgery under elective general anesthesia.

DETAILED DESCRIPTION:
Anatomical studies show that the 0.2% methylene blue was injected into the upper and lower surface of the gastrocnemius muscle and then diffused to the periphery.The common peroneal nerve, the medial sural cutaneous nerve, the lateral sural cutaneous nerve and the tibial nerve below the gastrocnemius muscle are all strongly stained (3 / 4 color of the nerve) or fully stained.

Previous clinical studies have shown that a single gastrocnemius muscle plane block can provide good postoperative analgesia after 16 hours for patients with foot and ankle surgery, significantly reduce the dose of opioids, and see no nerve injury.

Therefore, the investigators hypothesized that continuous gastrocnemius plane block could provide more lasting analgesia in patients undergoing foot-ankle surgery.

This clinical study uses a single-center, randomized, single-blind, parallel controlled trial design, divided into screening period, treatment period and follow-up periods.

Patients were randomized into two groups, the ropivacaine group and the control group.The venous access was open after home invasion and was routinely monitored electrocardiogram(ECG), non-invasive blood pressure(NBP) ，oxygen saturation(SpO2)，bispectral index(BIS). General anesthesia was performed.

Induction of anesthesia: propofol 1 milligram / kg, cis atracurium 0.2 milligrams / kilogram, sufentanil 10 micrograms ,remifentanil at 1.5 micrograms/ kilogram. Anesthesia maintenance: Propofol and sevoflurane static aspiration compound bispectral index was maintained at 40~60, remifentanil 0.3~0.4 μg / kg/min intravenous pump, and additional cis atracurium was added according to neuromuscular monitoring. In the postoperative ropivacaine group, the patient took a lateral decubitus position, and underwent a gastrocnemius plane block and catheterization under ultrasound guidance to connect a disposable electron infusion pump. (Formula of 0.125% ropivacaine of 300 milliliters, background dose of 3.0 milliliters / hour, patient controlled analgesia(PCA) dose of 8 milliliters , and locking time of 25 minutes). The control group received intravenous oxycodone titrated according to the numerical rating scale (NRS) score, and received no background dose of oxycodone patient-controlled intravenous analgesia (PCIA) pump for analgesia (single dose 1milligram, locking time 5minutes, 4 hours limit 12milligrams). All patients were given 50 milligrams of fluorophenol ester intravenously. Remedial analgesia: if patient controlled analgesia still can not tolerate the pain and numerical rating scale(NRS) ≥4, can be given intravenously oxycodone was done 2milligrams, separated by over 3 minutes, until numerical rating scale(NRS) ≤3.

Record: block range of 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 1 hour, 4 hours, 8 hours, 12 hours, 24 hours, 48hours and numerical rating scale(NRS) score during rest and exercise; time of first pressing of the analgesic pump; times of controlled analgesia (PCA); 0-4 hours, 0-8 hours, 0-16 hours, 0-24 hours, 8-16 hours, 16-24 hours, 24-32 hours, 32-40 hours,40-48 hours pain intensity-time curve (AUC); dose and times of remedial analgesic administration; Records: affected limb muscle strength and paresthesia, length of hospitalization, time of first ambulation, nausea and vomiting, neurological complications, patient satisfaction, physician and nurse satisfaction, etc.

The patient had open venous access after home invasion and was routinely monitored for electrocardiogram(ECG), non-invasive blood pressure(NBP) ，oxygen saturation(SpO2) and bispectral index(BIS). Induction and maintenance were performed according to a uniform anesthesia protocol. Postoperatively, the block was performed by the same anesthesiologist familiar with the ultrasound-guided nerve block. Various study indicators and data were collected by the same anesthesiologist who was not aware of the grouping situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective foot and ankle surgery
* Patient informed consent was obtained
* Age 18 to 65 years Sex is not limited
* American Society of Anesthesiologists(ASA)Ⅰ~Ⅲ level
* Body Mass Index(BMI)18~28kg/m2

Exclusion Criteria:

* Puncture site infection
* Abnormal coagulation function
* Local anesthetic allergy
* Severe cardiopulmonary disease
* Liver and renal insufficiency
* Medical history of chronic pain
* Long-term use of sedative and analgesic drugs
* Communication disorders
* The operation time exceeded 3 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-14 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Area under the pain intensity-time curve | Up to 48 hours postoperative
  The smaller the area under the pain intensity-time curve, the better the nerve block effect

SECONDARY OUTCOMES:
Percentage of subjects without remedial analgesics | Up to 48 hours postoperative
  The greater the percentage of subjects without remedial analgesics, the better the nerve block
The cumulative amount of remedial analgesic drugs (oxycodone) used | Up to 48 hours postoperative
  The smaller the cumulative amount of remedial analgesic drugs, the better the nerve blockade
Number of remedial analgesia | Up to 48 hours postoperative
  The less the remedial analgesia is, the better the nerve blockade is
Number of effective patient controlled analgesia (PCA) compressions | Up to 48 hours postoperative
  Number of effective patient controlled analgesia (PCA) compressions
The proportion of the number of invalid presses to the total presses | Up to 48 hours postoperative
  A smaller proportion of ineffective presses to total presses indicates a better nerve block
Total number of patient controlled analgesia (PCA) presses | Up to 48 hours postoperative
  Total number of patient controlled analgesia (PCA) presses

OTHER OUTCOMES:
The incidence of muscle strength and sensory abnormalities in the affected limb | Up to 48 hours postoperative
  The lower the incidence of muscle strength and sensory abnormalities in the affected limb, the better the effect of continuous gastrocnemius plane block
The incidence of adverse reactions, such as nausea, vomiting, and neurological complications | Up to 48 hours postoperative
  The lower the incidence of adverse effects such as nausea, vomiting, and neurological complications, the better the continuous gastrocnemius plane block technique
First time to get out of bed | Up to 48 hours postoperative
  First bedtime helps to judge the effect of the nerve block
The incidence of adverse events | Up to 48 hours postoperative
  Prevent adverse events such as catheter leakage and shedding
Patient satisfaction score | Up to 48 hours postoperative
  Rated on a 0-10 scale, with a higher score representing greater satisfaction.
The incidence of outbreak pain | Up to 7 days postoperative
  Patients with a single nerve block will have a burst of pain phenomenon, so we need to record the presence of a postoperative burst of pain phenomenon in patients with consecutive blocks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Provenzano DA, Viscusi ER, Adams SB Jr, Kerner MB, Torjman MC, Abidi NA. Safety and efficacy of the popliteal fossa nerve block when utilized for foot and ankle surgery. Foot Ankle Int. 2002 May;23(5):394-9. doi: 10.1177/107110070202300504. PMID 12043982
- [Background] Sun Li, Wei Jinju. Patient VAS was scored by ultrasound-guided continuous sciatic nerve block during foot surgery And the effect analysis of morphine dosage. Journal of Mathematical Medicine, 2019,32 (4): 523-524.
- [Background] Anderson JG, Bohay DR, Maskill JD, Gadkari KP, Hearty TM, Braaksma W, Padley MA, Weaver KT. Complications After Popliteal Block for Foot and Ankle Surgery. Foot Ankle Int. 2015 Oct;36(10):1138-43. doi: 10.1177/1071100715589741. Epub 2015 Jun 24. PMID 26109605
- [Background] Zhang Jinfang, Li Yimei. Ultrasound-guided continuous popliteal sciatic nerve block for postoperative analgesia in patients undergoing foot and ankle surgery. The World's Latest Medical Information Abstract, 2019,19 (68): 1-3.
- [Background] Qiu Wen, Yu Bin. Randomized controlled study of continuous popliteal sciatic nerve block analgesia and intravenous analgesia after foot and ankle surgery. Journal of Tongji University (Medical edition), 2 018,39 (02): 99-102.
- [Background] Gartke K, Portner O, Taljaard M. Neuropathic symptoms following continuous popliteal block after foot and ankle surgery. Foot Ankle Int. 2012 Apr;33(4):267-74. doi: 10.3113/FAI.2012.0267. PMID 22735198
- [Background] Bai Shu order, should be dajun et al. descriptive anatomy. The People's Health Publishing House. 353-357.
- [Background] Dong Guangyu, Huang Bingzhe, Zhang Hanyang, Chang Fei. Ankle joint block treatment. The Electronic Journal of Foot and Ankle Surgery. 2017, 4(3):59.

DOCUMENTS (1):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT05463809/Prot_000.pdf